CLINICAL TRIAL: NCT01086423
Title: Immunogenicity and Safety of GlaxoSmithKline Biologicals' DTPa-IPV/Hib (Infanrix-IPV+Hib™) in Infants
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Infanrix-IPV+Hib™ Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112584
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Tetanus; Poliomyelitis; Acellular Pertussis; Diphtheria; Haemophilus Influenzae Type b
Keywords: Infanrix-IPV+Hib
MeSH Terms: conditions — Tetanus; Poliomyelitis; Diphtheria; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (3):
- INFANRIX-IPV+HIB 1 GROUP (Experimental): Healthy male or female infants, between and including 60 and 90 days of age at the time of the first study visit, received 3 doses of Infanrix™-IPV+Hib vaccine at 2, 3 and 4 months of age, administered intramuscularly in the upper side of the right thigh.
  Interventions: Biological: Infanrix-IPV/Hib™
- INFANRIX-IPV+HIB 2 GROUP (Experimental): Healthy male or female infants, between and including 60 and 90 days of age at the time of the first study visit, received 3 doses of Infanrix™-IPV+Hib vaccine at 3, 4 and 5 months of age, administered intramuscularly in the upper side of the right thigh.
  Interventions: Biological: Infanrix-IPV/Hib™
- INFANRIX-HIB+POLIORIX GROUP (Active Comparator): Healthy male or female infants, between and including 60 and 90 days of age at the time of the first study visit, received 3 doses of Infanrix™-Hib vaccine co-administered with Poliorix™ vaccine at 2, 3 and 4 months of age, administered intramuscularly in the upper side of the right or left thigh, respectively.
  Interventions: Biological: Infanrix Hib™; Biological: Poliorix™

INTERVENTIONS:
Biological: Infanrix-IPV/Hib™ — Intramuscular, three doses
  Arms: INFANRIX-IPV+HIB 1 GROUP; INFANRIX-IPV+HIB 2 GROUP
Biological: Infanrix Hib™ — Intramuscular, three doses
  Arms: INFANRIX-HIB+POLIORIX GROUP
Biological: Poliorix™ — Intramuscular, three doses
  Arms: INFANRIX-HIB+POLIORIX GROUP

SUMMARY:
The purpose of the study is to evaluate the immunogenicity and reactogenicity of Infanrix-IPV/Hib™ vaccine when administered to healthy Chinese infants at 2, 3 and 4 or 3, 4 and 5 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between, and including, 60 and 90 days of age at the time of the first study visit.
* Born after a gestation period of 36 to 42 weeks, inclusive.
* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s) or LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Child in care.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period, with the exception of hepatitis B vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, poliomyelitis and/or Haemophilus influenzae type b (Hib) disease or vaccination.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.

The following condition is temporary or self-limiting and a subject may be vaccinated once the condition has resolved and no other exclusion criteria are met:

• Current febrile illness or axillary temperature > 37.0°C or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 985 (Actual)
Dates: Start 2010-03-01; Primary Completion 2010-11-19 (Actual); Study Completion 2010-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wuzhou, Guangxi, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 985 subjects originally enrolled in the study, 984 subjects were vaccinated with at least one dose of the study vaccine.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Infanrix-IPV+Hib 1 Group: Healthy male or female infants, between and including 60 and 90 days of age at the time of the first study visit, received 3 doses of Infanrix-IPV+Hib vaccine at 2, 3 and 4 months of age, administered intramuscularly in the upper side of the right thigh.
- Infanrix-IPV+Hib 2 Group: Healthy male or female infants, between and including 60 and 90 days of age at the time of the first study visit, received 3 doses of Infanrix-IPV+Hib vaccine at 3, 4 and 5 months of age, administered intramuscularly in the upper side of the right thigh.
- Infanrix-Hib+Poliorix Group: Healthy male or female infants, between and including 60 and 90 days of age at the time of the first study visit, received 3 doses of Infanrix-Hib vaccine co-administered with Poliorix vaccine at 2, 3 and 4 months of age, administered intramuscularly in the upper side of the right or left thigh, respectively.
Period: Overall Study
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Started | 330 | 324 | 330
Completed | 320 | 321 | 321
Not Completed | 10 | 3 | 9
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Migrated/moved from study area | 2 | 0 | 4
Not completed — Adverse event, fatal | 1 | 1 | 0
Not completed — Adverse event, non-fatal | 2 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group | Total
Number analyzed (Participants) | 330 | 324 | 330 | 984
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.9 (1.12) | 14.3 (1.14) | 9.9 (1.17) | 11.35 (2.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 147 | 141 | 443
  Male | 175 | 177 | 189 | 541
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Chinese heritage | 330 | 324 | 330 | 984

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphtheria (D) and Tetanus (T) Antigens
Description: A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: One month after the third vaccine dose (Month 3 or Month 4)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included a subset of evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against at least one study vaccine antigen component were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 147 | 156 | 147
Participants
  Anti-D | 146 | 156 | 147
  Anti-T | 147 | 156 | 147
Statistical Analysis 1: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™ -IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-D, one month after the third vaccine dose; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The upper limit (UL) of the standardized asymptotic 95% confidence interval (CI) on the group difference [Infanrix-Hib + Poliorix Group minus Infanrix-IPV+Hib 1 Group] in percentage of seroprotected subjects ≤ 10%; Difference in seroprotection rate = 0.68, 95% CI 2-sided [-1.88 to 3.76]
Statistical Analysis 2: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™-IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-T, one month after the third vaccine dose; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% CI on the group difference [Infanrix-Hib + Poliorix Group minus Infanrix-IPV+Hib 1 Group] in percentage of seroprotected subjects ≤ 10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.56 to 2.56]

2. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol-phosphate (PRP) Antigen
Description: A seroprotected subject was defined as a subject with anti-PRP antibody concentrations ≥ 0.15 micrograms per milliliter (μg/mL).
Time Frame: One month after the third vaccine dose (Month 3 or Month 4)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included a subset of evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against at least one study vaccine antigen component were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 147 | 157 | 150
Participants | 142 | 155 | 133
Statistical Analysis 1: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™-IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-PRP antibodies, one month after the third vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in seroprotection rate = -7.93, 95% CI 2-sided [-14.44 to -2.13]

3. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus Types 1, 2 and 3 Antigens
Description: A seroprotected subject was defined as a subject with anti-poliovirus (anti-polio) types 1, 2 and 3 antibody titres ≥ the value of 8.
Time Frame: One month after the third vaccine dose (Month 3 or Month 4)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 147 | 157 | 150
Participants
  Anti-polio 1 | 147 | 157 | 150
  Anti-polio 2 | 147 | 157 | 150
  Anti-polio 3 | 147 | 157 | 150
Statistical Analysis 1: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™-IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-Polio type 1 antibodies, one month after the third vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.51 to 2.56]
Statistical Analysis 2: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™-IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-Polio type 2 antibodies, one month after the third vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.51 to 2.56]
Statistical Analysis 3: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™-IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-Polio type 3 antibodies, one month after the third vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.51 to 2.56]

4. Primary Outcome: Number of Subjects With a Vaccine Response to Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) Antigens
Description: Vaccine response was defined as:
  For PT and FHA response, antibody concentration ≥ 20 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL) at post-vaccination.
  For PRN response: for initially seronegative subjects [antibody concentration lower than (<) 5 EL.U/mL], post-vaccination antibody concentration ≥ 20 EL.U/mL; for initially seropositive subjects (antibody concentration ≥ 5 EL.U/mL), at least a 4-fold increase in antibody concentration from pre to post-vaccination.
Time Frame: One month after the third vaccine dose (Month 3 or Month 4)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 147 | 156 | 148
Participants
  Anti-PT | 147 | 155 | 147
  Anti-FHA | 147 | 155 | 144
  Anti-PRN | 145 | 156 | 145
Statistical Analysis 1: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™-IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-PT antigens, one month after the third vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in seroprotection rate = -0.68, 95% CI 2-sided [-3.74 to 1.89]
Statistical Analysis 2: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™-IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-FHA antigens, one month after the third vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in seroprotection rate = -2.7, 95% CI 2-sided [-6.75 to -0.11]
Statistical Analysis 3: Comparison: Infanrix-IPV+Hib 1 Group vs Infanrix-Hib+Poliorix Group; To demonstrate that the immunogenicity of Infanrix™-IPV+Hib vaccine administered at 2, 3 and 4 months of age was non-inferior to that of the concomitant administration of Infanrix™-Hib and Poliorix™ vaccines at the same age, in terms of immune response to anti-PRN antigens, one month after the third vaccine dose; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: The UL of the standardized asymptotic 95% confidence interval (CI) on the group difference [Infanrix-Hib + Poliorix Group minus Infanrix-IPV+Hib 1 Group] in percentage of seroprotected subjects ≤ 10%; Difference in seroprotection rate = -0.67, 95% CI 2-sided [-4.6 to 3.04]

5. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in IU/mL.
Time Frame: Before the first dose (Month 0) and one month after the third dose of vaccination (Month 3 or Month 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 147 | 157 | 151
IU/mL
  Anti-D, M0 | 0.052 [0.05 to 0.053] | 0.051 [0.05 to 0.052] | 0.051 [0.049 to 0.052]
  Anti-D, M3/M4: number analyzed (Participants) | 147 | 156 | 147
  Anti-D, M3/M4 | 0.719 [0.661 to 0.782] | 0.753 [0.699 to 0.812] | 0.613 [0.565 to 0.666]
  Anti-T, M0 | 0.051 [0.05 to 0.052] | 0.052 [0.05 to 0.054] | 0.05 [0.05 to 0.05]
  Anti-T, M3/M4: number analyzed (Participants) | 147 | 156 | 147
  Anti-T, M3/M4 | 4.118 [3.779 to 4.488] | 4.124 [3.796 to 4.479] | 3.618 [3.339 to 3.921]

6. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in µg/mL.
Time Frame: Before the first dose (Month 0) and one month after the third dose of study vaccine (Month 3 or Month 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 147 | 157 | 151
µg/mL
  Anti-PRP, M0: number analyzed (Participants) | 146 | 157 | 151
  Anti-PRP, M0 | 0.127 [0.104 to 0.154] | 0.135 [0.112 to 0.163] | 0.15 [0.122 to 0.185]
  Anti-PRP, M3/M4: number analyzed (Participants) | 147 | 157 | 150
  Anti-PRP, M3/M4 | 5.601 [4.676 to 6.709] | 9.396 [8.032 to 10.992] | 2.826 [2.235 to 3.572]

7. Secondary Outcome: Anti-polio Types 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Before the first dose (Month 0) and one month after the third dose of study vaccine (Month 3 or Month 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 147 | 157 | 151
Titers
  Anti-polio 1, M0: number analyzed (Participants) | 146 | 157 | 151
  Anti-polio 1, M0 | 9.4 [7.7 to 11.5] | 7.1 [6.2 to 8.2] | 9.2 [7.7 to 11]
  Anti-polio 1, M3/M4: number analyzed (Participants) | 147 | 157 | 150
  Anti-polio 1, M3/M4 | 1143.7 [952.7 to 1372.9] | 1328.9 [1137.6 to 1552.4] | 533.6 [469.5 to 606.4]
  Anti-polio 2, M0: number analyzed (Participants) | 146 | 157 | 151
  Anti-polio 2, M0 | 6.3 [5.5 to 7.2] | 5 [4.6 to 5.5] | 6.9 [6 to 8]
  Anti-polio 2, M3/M4: number analyzed (Participants) | 147 | 157 | 150
  Anti-polio 2, M3/M4 | 416.2 [344.5 to 502.8] | 458.6 [385.6 to 545.5] | 186.4 [160.4 to 216.5]
  Anti-polio 3, M0: number analyzed (Participants) | 146 | 157 | 151
  Anti-polio 3, M0 | 5.8 [5 to 6.8] | 4.9 [4.3 to 5.6] | 5.7 [5.1 to 6.4]
  Anti-polio 3, M3/M4: number analyzed (Participants) | 147 | 157 | 150
  Anti-polio 3, M3/M4 | 1478.8 [1210.6 to 1806.5] | 1411.6 [1175.3 to 1695.3] | 820.7 [820.7 to 964.4]

8. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: Before (Month 0) and one month after the third dose of study vaccine (Month 3 or Month 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 147 | 157 | 151
EL.U/mL
  Anti-PT, M0 | 2.9 [2.8 to 3.1] | 2.7 [2.6 to 2.8] | 2.8 [2.6 to 2.9]
  Anti-PT, M3/M4: number analyzed (Participants) | 147 | 156 | 148
  Anti-PT, M3/M4 | 108.7 [99.2 to 119.1] | 114.7 [105.4 to 124.8] | 97.1 [88.3 to 106.8]
  Anti-FHA, M0 | 2.9 [2.7 to 3.1] | 2.6 [2.5 to 2.7] | 2.9 [2.7 to 3.1]
  Anti-FHA, M3/M4: number analyzed (Participants) | 147 | 156 | 148
  Anti-FHA, M3/M4 | 87.7 [79.9 to 96.3] | 87.6 [79.6 to 96.4] | 76.3 [68.5 to 85]
  Anti-PRN, M0 | 2.6 [2.5 to 2.7] | 2.6 [2.5 to 2.6] | 2.5 [2.5 to 2.6]
  Anti-PRN, M3/M4: number analyzed (Participants) | 147 | 156 | 148
  Anti-PRN, M3/M4 | 44.8 [42 to 47.9] | 43.7 [41.3 to 46.3] | 43.2 [39.8 to 47]

9. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 330 | 324 | 330
Participants
  Any Pain, Dose 1 | 65 | 64 | 83
  Any Redness, Dose 1 | 16 | 19 | 15
  Any Swelling, Dose 1 | 8 | 9 | 9
  Any Pain, Dose 2: number analyzed (Participants) | 321 | 321 | 322
  Any Pain, Dose 2 | 43 | 50 | 58
  Any Redness, Dose 2: number analyzed (Participants) | 321 | 321 | 322
  Any Redness, Dose 2 | 14 | 19 | 13
  Any Swelling, Dose 2: number analyzed (Participants) | 321 | 321 | 322
  Any Swelling, Dose 2 | 6 | 8 | 8
  Any Pain, Dose 3: number analyzed (Participants) | 321 | 321 | 321
  Any Pain, Dose 3 | 39 | 41 | 39
  Any Redness, Dose 3: number analyzed (Participants) | 321 | 321 | 321
  Any Redness, Dose 3 | 10 | 11 | 8
  Any Swelling, Dose 3: number analyzed (Participants) | 321 | 321 | 321
  Any Swelling, Dose 3 | 5 | 8 | 6
  Any Pain, Across doses | 90 | 91 | 102
  Any Redness, Across doses | 28 | 34 | 26
  Any Swelling, Across doses | 14 | 17 | 19

10. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above 37.0 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relationship to study vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period after each vaccine dose and across doses
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 330 | 324 | 330
Participants
  Any Drowsiness, Dose 1 | 95 | 80 | 69
  Any Irritability, Dose 1 | 123 | 120 | 116
  Any Loss of appetite, Dose 1 | 77 | 86 | 76
  Any Fever/Axillary, Dose 1 | 137 | 152 | 103
  Any Drowsiness, Dose 2: number analyzed (Participants) | 321 | 321 | 322
  Any Drowsiness, Dose 2 | 53 | 47 | 53
  Any Irritability, Dose 2: number analyzed (Participants) | 321 | 321 | 322
  Any Irritability, Dose 2 | 96 | 100 | 103
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 321 | 321 | 322
  Any Loss of appetite, Dose 2 | 69 | 72 | 59
  Any Fever/Axillary, Dose 2: number analyzed (Participants) | 321 | 321 | 322
  Any Fever/Axillary, Dose 2 | 131 | 144 | 102
  Any Drowsiness, Dose 3: number analyzed (Participants) | 321 | 321 | 321
  Any Drowsiness, Dose 3 | 43 | 32 | 28
  Any Irritability, Dose 3: number analyzed (Participants) | 321 | 321 | 321
  Any Irritability, Dose 3 | 77 | 70 | 61
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 321 | 321 | 321
  Any Loss of appetite, Dose 3 | 65 | 57 | 36
  Any Fever/Axillary, Dose 3: number analyzed (Participants) | 321 | 321 | 321
  Any Fever/Axillary, Dose 3 | 93 | 82 | 75
  Any Drowsiness, Across doses | 124 | 102 | 99
  Any Irritability, Across doses | 171 | 166 | 163
  Any Loss of appetite, Across doses | 131 | 136 | 114
  Any Fever/Axillary, Across doses | 217 | 217 | 183

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period after any dose
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 330 | 324 | 330
Participants | 98 | 114 | 110

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 to Month 4/5)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
Number analyzed (Participants) | 330 | 324 | 330
Participants | 6 | 3 | 4

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period. Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period. SAEs: during the entire study period (from Month 0 up to Month 4/5).
Arm/Group | Infanrix-IPV+Hib 1 Group | Infanrix-IPV+Hib 2 Group | Infanrix-Hib+Poliorix Group
All-Cause Mortality (participants affected / at risk) | 1/330 | 0/324 | 0/330
Serious Adverse Events (participants affected / at risk) | 6/330 | 3/324 | 4/330
Other Adverse Events (participants affected / at risk) | 279/330 | 277/324 | 272/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV+Hib 1 Group (N=330) | Infanrix-IPV+Hib 2 Group (N=324) | Infanrix-Hib+Poliorix Group (N=330)
Enteritis (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Hepatitis neonatal (Hepatobiliary disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 3 | 2 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV+Hib 1 Group (N=330) | Infanrix-IPV+Hib 2 Group (N=324) | Infanrix-Hib+Poliorix Group (N=330)
Pyrexia (General disorders) | 19 | 24 | 17
Pain (General disorders) | 90 | 91 | 102
Redness (General disorders) | 28 | 34 | 26
Swelling (General disorders) | 14 | 17 | 19
Drowsiness (General disorders) | 124 | 102 | 99
Irritability (General disorders) | 171 | 166 | 163
Loss of appetite (General disorders) | 131 | 136 | 114
Fever (Axillary) (General disorders) | 217 | 217 | 183
Diarrhoea (Gastrointestinal disorders) | 23 | 22 | 33
Nasopharyngitis (General disorders) | 42 | 46 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.